CLINICAL TRIAL: NCT05277610
Title: Iron Status and Its Relation to Lung Function in Pediatric Asthmatics
Brief Title: Iron Status and Lung Function in Pediatric Asthma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba Omara, DR. Heba omara, Ain Shams University
Other Study IDs: AinShamsU555
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Function Tests
Keywords: asthma, pediatric, iron deficiency anemia
MeSH Terms: conditions — Asthma; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: iron studies — Pulmonary function testing was performed using standardized spirometry for asthmatic patients with iron deficiency anemia and those without iron deficiency anemia

SUMMARY:
Iron has a variable role regarding asthma and respiratory function. In addition, iron deficiency may affect spirometry results in asthmatic children. So, we aimed to assess the effect of ion status on lung function in childhood asthma

DETAILED DESCRIPTION:
This cross-sectional study included fifty asthmatic children in the age group of 6-16 years. Asthmatic patients were classified according to their complete blood count and iron profile into 2 groups: group 1; asthmatic children without iron deficiency anemia (IDA), group 2; asthmatic children with IDA. All patients underwent full history taking, clinical examination, laboratory investigations, asthma control test, and pulmonary function tests.

Pulmonary function testing was performed using standardized spirometry. Lung function was measured by forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC, and maximal mid-expiratory flow (MMEF 25-75%) of FVC. both patients' groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of bronchial asthma: The diagnosis of bronchial asthma in the studied children was based on clinical examination The diagnosis of iron deficiency anemia was supported by criteria provided and updated by the World Health Organization

Exclusion Criteria:

* chronic lung diseases other than asthma Severe systemic illnesses such as liver, renal diseases, and nutritional disorders

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Asthmatic children with and without iron deficiency anemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
improved asthma control | 2 months
  higher asthma control test

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Omara, Cairo, Lecturer/Instructor, Egypt

IPD SHARING:
Plan to Share IPD: No